CLINICAL TRIAL: NCT05390827
Title: Remote Digital Physiological Data Collection in Cancer: An MSK Registry Protocol
Brief Title: Remote Digital Physiologic Data Collection in Cancer: An MSK Registry Protocol
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-330
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor
Keywords: Remote Digital Physiological Data Collection; Exercise Oncology; 20-330

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a secure method of collecting physiologic information from patients with cancer. The researchers will use this information to learn more about how physiologic data may relate to cancer diagnosis and response to treatment, and to identify factors that may lead to higher or lower risk of cancer.

DETAILED DESCRIPTION:
Project 1: HealthKit This prospective registry cohort study will aim to recruit a total of 3,000 patients and 500 adults without a history of cancer. The targeted patient cohorts / settings will aim to be : (1) pre-treatment / during treatment: patients with newly diagnosed early-stage, low-grade, or locally advanced solid tumors that are either pre- or during treatment, (2) post-treatment: patients with primary solid tumor diagnose is that are post-treatment, (3) advanced disease setting: patients diagnosed with metastatic or high-grade disease, (4) patients enrolled onto investigational trials in the early drug development (EDD) Service, (5) patients admitted to Urgent Care Center (UCC), and (6) patients completing a Survivorship Patient Self-Assessment as part of follow-up in an MSK Survivorship clinic. This study will accrue patients receiving care at any MSK site. Adults without a history of cancer will be recruited as a comparison group. The targeted adults without a history of cancer cohorts will aim to be (n=250/cohort): (7) adults without a history of cancer <50 years of age, and (8) adults without a history of cancer aged greater than or equal to 50 years.

Project 2: DigIT-Ex This prospective registry cohort study will aim to recruit a total of 120 patients and 24 adults without a history of cancer. The targeted adult patient cohorts / settings will be (n=12/cohort), excluding cohort 6, which will be (n=48): (1) patients scheduled to undergo bone marrow transplantation, (2) patients newly diagnosed with acute myeloid leukemia (AML), (3) patients scheduled to undergo surgery for localized prostate cancer (4) patients scheduled to undergo surgery for lung cancer, (5) patients scheduled to undergo total neoadjuvant therapy for advanced rectal cancer, (6) patients scheduled to undergo antiandrogen therapy for advanced prostate cancer, and (7) patients scheduled to undergo chemotherapy for metastatic pancreatic cancer. The targeted adults without a history of cancer cohorts will be (n=12/cohort): (8) individuals without a history of cancer aged less than 50 years, and (9) individuals without a history of cancer aged greater than or equal to 50 years.

ELIGIBILITY:
Inclusion Criteria:

Project 1: HealthKit

* Individuals who meet at least one of the following criteria:

  * Diagnosis of new onset early-stage (I-III), low-grade (I-II), or locally advanced solid tumor
  * Historical diagnosis of primary invasive solid tumor
  * Diagnosis of metastatic (stage IV) or high-grade (III-IV) disease
  * Enrolled onto an investigational trial in the EDD Service
  * Seen in the MSK UCC from 2021 and onwards
  * Completion of Survivorship Patient Self-Assessment
  * Adult without a history of cancer <50 years of age
  * Adult without a history of cancer ≥ 50 years of age
* ≥18 years old
* Own an Apple iPhone with valid iOS operating software
* Have a registered MSK MyChart account and be willing to download the MSK Remote Monitoring (RM) application onto their personal iPhone
* Self-reported "very well" comprehension of written and verbal English language
* Willing and able to provide informed consent and HIPAA authorization for the release of personal health information

Project 2: DigIT-Ex

Individuals who meet one of the following criteria:

* Patients at MSK who are:
* Scheduled to undergo any type of BMT (Cohort 1)
* Diagnosed with new onset AML and scheduled to initiate antineoplastic therapy (Cohort 2)
* Scheduled to undergo any surgery for prostate cancer (Cohort 3)
* Scheduled to undergo any lung cancer surgery (Cohort 4)
* Scheduled to undergo TNT for locally advanced rectal cancer (Cohort 5)
* Scheduled to initiate androgen deprivation therapy for at least 12 months and has one of the following prostate cancer diagnoses (Cohort 6):
* High risk/very high localized, locally advanced,
* Biochemically recurrent prostate cancer
* Treatment naïve, low-volume metastatic prostate cancer
* Scheduled Scheduled to undergo chemotherapy for metastatic pancreatic cancer (Cohort 7)
* Individuals without cancer <50 years of age (Cohort 8)
* Individuals without cancer ≥50 years of age (Cohort 9)

  * 18 to 90 years old at the time of consent
  * Willing and able to download the Withings Health Mate app onto their personal mobile device
  * Willing to provide mobile digital physiological data for a period of at least six months to a maximum of one year following consent
  * Willing to provide informed consent

Exclusion Criteria:

Project 1: HealthKit

* Unable or unwilling to successfully export and /or share physiological data

Project 2: DigIT-Ex

* Unable or unwilling to appropriately use digital platforms or devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified by a member of the patient's care team, a protocol investigator, or research staff at Memorial Sloan Kettering Cancer Center (MSK).
Sampling Method: Non-Probability Sample
Enrollment: 3644 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
establish a mechanism within the institution to prospectively collect / extract digital remote physiological data among patients with cancer | 1 year
  to create a repository and infrastructure to address novel questions of clinical importance.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Pike, MD, DPhil, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm